CLINICAL TRIAL: NCT01770171
Title: A Randomized Phase II Trial of Carboplatin-Paclitaxel Compared to Carboplatin-Paclitaxel-Bevacizumab in Advanced (Stage III-IV) or Recurrent Endometrial Cancer
Brief Title: Carboplatin-Paclitaxel ± Bevacizumab in Advanced (Stage III-IV) or Recurrent Endometrial Cancer
Acronym: MITOBEVAEND2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor Giovanni Scambia, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITOBEVAEND2
Record Dates: First submitted 2012-12-10; First posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2012-12

CONDITIONS: Stage III-IV or Recurrent Endometrial Cancer
Keywords: endometrial cancer; recurrent endometrial cancer; bevacizumab
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin-paclitaxel-bevacizumab (Experimental): Carboplatin AUC 5+ Paclitaxel 175 mg/mq+Bevacizumab 15 mg/kg q 21 for 6 -8 cycles + Bevacizumab 15 mg/kg every 3 weeks until disease progression
  Interventions: Drug: Bevacizumab
- carboplatin-paclitaxel (Active Comparator): Carboplatin AUC 5+Paclitaxel 175 mg/mq q 21 for 6-8 cycles
  Interventions: Drug: Carboplatin AUC 5+Paclitaxel 175 mg/mq q 21 for 6-8 cycles

INTERVENTIONS:
Drug: Bevacizumab — Carboplatin AUC 5+ Paclitaxel 175 mg/mq+Bevacizumab 15 mg/kg q 21 for 6 -8 cycles + Bevacizumab 15 mg/kg
  Arms: Carboplatin-paclitaxel-bevacizumab
Drug: Carboplatin AUC 5+Paclitaxel 175 mg/mq q 21 for 6-8 cycles — Carboplatin AUC 5+Paclitaxel 175 mg/mq q 21 for 6-8 cycles
  Arms: carboplatin-paclitaxel

SUMMARY:
Wright et al (Anticancer Res, 2000) reported the results of a retrospective study on 11 patients with advanced/recurrent endometrial cancers. All patients had multi-site disease and were heavily pretreated with a median of 3 prior chemotherapy regimens. All received bevacizumab combination therapy which was well-tolerated. Two patients had partial responses, 3 had stable disease, while 5 patients progressed. One subject was not assessable for response. The median progression-free interval was 5.4 months for the entire cohort and 8.7 months for those who achieved clinical benefit (PR or SD). The authors concluded that Bevacizumab was well-tolerated and displayed promising anti-neoplastic activity in patients with endometrial cancer.The rationale for combining anti-angiogenic agents, including anti-VEGF antibodies, with cytotoxic chemotherapy stems from a number of preclinical studies showing additive and synergistic anti-tumour activity in a number of solid tumour types. By combining VEGF-targeting agents such as bevacizumab with conventional chemotherapies, it is hoped that these agents will act synergistically, thereby enhancing their anti-tumour efficacy and controlling disease progression.

The addition of bevacizumab to chemotherapy has been shown to improve PFS and/or OS in a series of large, randomized Phase III clinical trials in a wide range of tumour types, including mCRC, non-squamous NSCLC, metastatic BC (mBC) and mRCC.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. ECOG Performance Status of 0-2.
3. Life expectancy of at least 12 weeks.
4. Patients must have advanced stage III or IV, or recurrent histologically-confirmed endometrial cancer.
5. Endometrial cancer will include all carcinomas, including endometrioid carcinoma, papillary serous carcinoma, clear cell carcinoma.
6. One previous chemotherapy lines is allowed if platinum free interval is more than six mounths (previous radiotherapy is allowed).

7 Measurable and not measurable disease. 8 Adequate renal and hepatic function, defined as:

* Total serum bilirubin ≤ institutional ULN unless patient has Gilbert's syndrome in which case direct bilirubin must be < ULN for the institution.
* AST and/or ALT ≤ 2.5 x ULN for the institution. (or ≤ 5 x ULN if liver metastases are present)
* Alkaline phosphatase < 1.5 x ULN for the institution (if > 1.5 x ULN, then alkaline phosphatase liver fraction must be < 1.5 ULN).
* Serum creatinine ≤ 1.5 x ULN for the institution (or calculated creatinine clearance ≥ 50 mL/min/1.73 m2) 9 Adequate bone marrow function, defined as:
* Total leukocytes ³ 3.0 x 109/L.
* ANC ³ 1.5 x 109/L.
* Platelet count ³ 100 x 109/L. Able to understand and give written informed consent. 10 Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

1. Previous cytotoxic chemotherapy.
2. Women who are pregnant or lactating.
3. Presence of brain or other central nervous system metastases.
4. Anticancer treatment within 4 weeks prior to randomization.
5. Ongoing toxicity associated with prior anticancer therapy.
6. Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 4 weeks prior to randomization. Patients who have recovered from placement of a central venous access port within 2 weeks of Cycle 1 Day 1 will be considered eligible.
7. Another primary malignancy within the past five years (except for non-melanoma skin cancer and cervical carcinoma in situ).
8. Current or recent (within 10 days prior to the first study drug dose) chronic daily treatment with aspirin (>325 mg/day).
9. Current or recent (within 10 days prior to the first study drug dose) use of full-dose oral or parenteral anticoagulant or thrombolytic agent for therapeutic purposes.
10. Inadequate coagulation parameters:activated partial thromboplastin time (APTT) >1.5 xULN or INR >1.5.
11. Known HIV infection.
12. Known hepatitis B or C infection.
13. Concurrent treatment with immunosuppressive or investigational agents.
14. History or evidence of thrombotic or hemorrhagic disorders; including cerebrovascular accident (CVA) / stroke or transient ischemic attack (TIA) or subarachnoid haemorrhage within _6 months prior to the first study treatment).
15. Uncontrolled hypertension (sustained systolic >150 mm Hg and/or diastolic >100 mm Hg despite antihypertensive therapy) or clinically significant (i.e. active) cardiovascular disease, including.
16. Myocardial infarction or unstable angina within _6 months prior to the first study treatment.
17. New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF).
18. Serious cardiac arrhythmia requiring medication (with the exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
19. Peripheral vascular disease _grade 3 (i.e.symptomatic and interfering with activities of daily living requiring repair or revision).
20. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to the first study treatment.
21. Non-healing wound, ulcer or bone fracture. Patients with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection are eligible but require three weekly wound examinations.
22. Serious active infection requiring i.v. antibiotics at enrolment.
23. Significant traumatic injury during the 4 weeks preceding the first dose of bevacizumab.
24. Known hypersensitivity to any of the study drugs or excipients (including cremophor and hamster Ovary cell products).
25. Evidence of any other medical conditions (such as psychiatric illness, peptic ulcer, etc.), physical examination or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment related complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2012-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 months
  • Progression-free survival, defined as the time from the date of randomization to the date of documented progressive disease, recurrence or death (whichever occurs first)

SECONDARY OUTCOMES:
Overall survival | 3 months
  • Overall survival defined as the time from the date of randomization to the date of death
Best target lesion response | 6 months
  Best target lesion response, defined as best change in sum of the target lesions from baseline to disease progression.
Duartion of Response | 3 months
  Duration of response Safety and tolerability
Quality of life | 3 cycle
  Changes Quality of Life parameters as measured using EORTC QLQ-30 & EORTC-QLQ-EN-24

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Prof, Principal Investigator — Catholic University of Sacred Heart; Domenica Lorusso, MD, Principal Investigator — National Cancer Institute, Milan
Locations (1):
- Catholic University of Sacred Heart Rome,, Rome, Rome, Italy